CLINICAL TRIAL: NCT04117581
Title: A Daily 5000 IU Vitamin D Supplement for the Improvement of Lung Function and Asthma Control in Adults With Asthma: a Randomised Controlled Trial
Brief Title: A Study to Investigate the Effect of Vitamin D3 Supplementation on Asthma Symptoms in Adults With Asthma (VITDAS)
Acronym: VITDAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1583/19/SW/CSN
Record Dates: First submitted 2019-10-04; First posted 2019-10-07 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-02

CONDITIONS: Asthma; Vitamin D Deficiency; Nutritional Deficiency; Inflammation
Keywords: Vitamin D; Asthma; Lung function; Inflammation
MeSH Terms: conditions — Asthma; Vitamin D Deficiency; Malnutrition; Inflammation | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D3 supplement (Active Comparator): Participant will be asked to take one capsule of vitamin D3 supplement (5000 IU) (125 μg) daily for a total duration of 12 weeks.
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): Participants will be asked to take one capsule of placebo (inert filler) daily for a total duration of 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 5000 IU (125 μg) vitamin D3 capsules daily over 12 weeks (84 days)
  Other Names: Cholecalciferol
  Arms: Vitamin D3 supplement
Other: Placebo — Inert filler capsules daily over 12 weeks (84 days)
  Other Names: Non active ingredient
  Arms: Placebo

SUMMARY:
Asthma is a disease characterised by chronic inflammation of the airways leading to symptoms including periods of shortness of breath, wheezing and a tight chest due to airway narrowing in affected patients. Current data show that one in 12 adults are currently receiving treatment for asthma in the United Kingdom (UK), with the UK having some of the highest rates in Europe. In the winter, 30-40% of the UK population are vitamin D deficient with some asthma patients having significantly lower vitamin D levels compared to normal patients. Vitamin D has been shown to be involved in the development of immune-related disorders including asthma. Cross-sectional research has shown that reduced vitamin D levels are associated with reduced lung function, increased airway hyper-responsiveness and reduced response to glucocorticoids, suggesting vitamin D levels may also implicate asthma treatment. To date, there have been three randomised controlled trials (RCT) assessing the effect of vitamin D supplementation in adults with symptomatic asthma. These trials have not found a significant effect of vitamin D supplementation on asthma. However, these studies relied on high doses of vitamin D with long time periods between doses. There is a requirement for RCTs in adults with daily supplementation of lower doses of vitamin D as it has been suggested that daily supplementation is more effective for inducing non-classical actions of vitamin D. However, vitamin D has been found to significantly improve airway function as measured by forced expiratory volume in one second (FEV1) in adults supplemented with 100, 000 international units (IU) vitamin D intramuscularly plus 50, 000 IU oral vitamin D weekly. Therefore, the effect of daily dosing on lung function also requires investigation. Furthermore, these trials have focussed on clinical outcomes without investigating the cellular mechanisms affording protection.

DETAILED DESCRIPTION:
Recruitment and sampling strategy:

Participants will be recruited from the University of Chester (staff and students) and surrounding areas, United Kingdom (UK) only. Emails, posters and social media will be used to advertise the study to the target group (adults with asthma). A total of 28 adults with asthma aged 18-65 years old will be included in the study based on criteria described below. Eligibility will be based upon previous diagnosis of asthma by a general practitioner (GP) and the number of times asthma medication is required at screening before the start of the study. Participants will be required to complete a screening questionnaire which will provide information about participant's health status, drugs/medication/supplement usage and sun exposure. Those that have had asthma diagnosed by a GP and require their medication more than twice per week will be included. All eligible participants will be briefed on the study protocol before the beginning of the study, and the eligible participants will be given a participant information sheet (PIS) and asked to provide written informed consent.

A 12 week, double blind, randomised controlled trial will be carried out in the clinical laboratory at The University of Chester, UK. Most vitamin D and asthma studies have used supplement concentrations up to 120, 000 international units (IU) with no adverse effects. The European Food Standards Agency (EFSA) set a no-observed-adverse-effect-level (NOAEL) of 10,000IU/day (COT, 2015).

Participants will be randomly allocated to 2 groups:

1. vitamin D group
2. placebo group

Participants assigned to the vitamin D group will consume one capsule containing 5000 IU vitamin D every day. Participants in the placebo group will take an identical capsule containing inert filler. Participants will be asked to maintain their dietary habits and physical activity. The remaining supplements will be returned at the final clinic (week 12) and compliance will be estimated.

Participants will be required to attend three clinics in total over a period of 12 weeks, and they will be assessed at baseline (Day 0), interim (Week 6) and post-intervention (Week 12). At each clinic, a 30ml blood sample will be taken and both height and weight will be measured. Before the start and end of the study, participants will be required to keep a 3-day food diary which includes two weekdays and one weekend day to represent the habitual dietary intake of the participants. At each clinic, participants will complete spirometry to measure forced expiratory volume in one second (FEV1) and forced vital capacity (FVC) to assess lung function and complete the Asthma Control Test™ (ACT) to assess asthma symptoms. Blood samples will be analysed on collection for a total blood cell count. Blood samples will be centrifuged to remove plasma. Plasma samples will be batch analysed at the end of the intervention to assess biomarkers of vitamin D metabolism and inflammation.

Sample size and justification:

Sample size was estimated using vitamin D supplementation data from a study in which FEV1 post intervention at 6 months (mean ± standard deviation (S.D)) of 51.6 ± 9.4 L (vitamin D treatment group) and 31.9 ± 7.6 L (placebo group) was reported in chronic obstructive pulmonary disease patients receiving 100, 000 IU vitamin D each month. With an effect size of 1.8493555, the total sample size required for each group in the proposed study is 9. Taking into account a 20% drop out rate, and this study lasting only 12 weeks, the total sample size required is 14 (power = 0.9). Therefore, the total sample size needed for the whole study is 28. Sample size was estimated using G Power Software.

Statistical Analysis:

All statistical analyses will be conducted with the International Business Machines (IBM) Statistical Package for the Social Sciences (SPSS) Statistic Data Editor Software (version 25). Assuming the data is normally distributed after performing a Shapiro Wilks normality test, a mixed model analysis of variance (ANOVA) with t-test post-hoc analysis will be conducted to compare the mean differences for all measured parameters between the groups at the different time points. A non-parametric approach will be adopted if the data is not normally distributed for all analyses. Differences will be considered significant with a p value ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 years to 65 years
2. Asthma diagnosed by a general practitioner
3. Taking inhaled therapy to treat asthma that is required at least two times per week

Exclusion Criteria:

1. Taking vitamin D supplements or supplements containing calcium
2. History of asthma requiring treatment with intubation and mechanical ventilation within the past five years
3. Require inhaled asthma therapy more than four times per day
4. Respiratory tract infection within the past four weeks
5. Suffering from chronic diseases of the lung (other than asthma), heart, liver, kidney, endocrine or nervous system or immunodeficiency
6. History of smoking within the past year or > 10 years total
7. Been on a sun holiday within a month of taking part in the study or during the study. For the purpose of this study a sun holiday is defined as: spending one week or more in a hotter climate with the intention of sun-bathing
8. Unable to communicate in English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change in lung function from baseline to 12 weeks | 0 weeks, 6 weeks, 12 weeks
  Forced expiratory volume in one second (FEV1) and forced expiratory volume (FVC) measured by spirometry

SECONDARY OUTCOMES:
Change in Asthma Control Test™ score | 0 weeks, 6 weeks, 12 weeks
  Indication of level of asthma control according to participant. Score between 0 and 25.
  Scores indicate:
  25: Asthma appears to have been under control over the last 4 weeks 20 - 24: Asthma appears to have been reasonably well controlled over the last 4 weeks Less than 20: Asthma may not have been controlled during the past 4 weeks
Change in vitamin D concentration from baseline to 12 weeks | 0 weeks, 6 weeks, 12 weeks
  Vitamin D3 status measured in plasma samples by enzyme-linked immunosorbent assay (ELISA) commercial kit
Change in parathyroid hormone (PTH) concentration from baseline to 12 weeks | 0 weeks, 6 weeks, 12 weeks
  Vitamin D metabolism biomarker measured in plasma samples by ELISA commercial kit
Change in Full Blood Count Concentration from baseline to 12 weeks | 0 weeks, 6 weeks, 12 weeks
  Percentage granulocytes measured in whole blood samples by Beckman Coulter haematological analyser
Change in interferon-gamma (IFN-ϒ) concentration from baseline to 12 weeks | 0 weeks, 6 weeks, 12 weeks
  Inflammatory biomarker measured in plasma samples by ELISA commercial kit
Change in tumour-necrosis-factor-alpha (TNF-α) concentration from baseline to 12 weeks | 0 weeks, 6 weeks, 12 weeks
  Inflammatory biomarker measured in plasma samples by ELISA commercial kit
Change in C-reactive protein (CRP) concentration from baseline to 12 weeks | 0 weeks, 6 weeks, 12 weeks
  Inflammatory biomarker measured in plasma samples by ELISA commercial kit
Change in immunoglobulin E (IgE) concentration from baseline to 12 weeks | 0 weeks, 6 weeks, 12 weeks
  Antibody measured in plasma samples by ELISA commercial kit
Change in interleukin-(IL)4 concentration from baseline to 12 weeks | 0 weeks, 6 weeks, 12 weeks
  Inflammatory biomarker measured in plasma samples by ELISA commercial kit
Change in IL-10 concentration from baseline to 12 weeks | 0 weeks, 6 weeks, 12 weeks
  Inflammatory biomarker measured in plasma samples by ELISA commercial kit
Change in IL-13 concentration from baseline to 12 weeks | 0 weeks, 6 weeks, 12 weeks
  Inflammatory biomarker measured in plasma samples by ELISA commercial kit

CONTACTS AND LOCATIONS:
Overall Officials: Sohail Mushtaq, PhD, Principal Investigator — University of Chester
Locations (1):
- University of Chester, Chester, Chesire, United Kingdom

IPD SHARING:
Plan to Share IPD: No